CLINICAL TRIAL: NCT06804057
Title: CorEvitas Systemic Lupus Erythematosus (SLE) Drug Safety and Effectiveness Registry
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-SLE-800
Record Dates: First submitted 2024-12-02; First posted 2025-01-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Peripheral blood for serum, plasma, DNA, and RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Collection — Blood will be collected for the subjects who are willing to participate in the optional biorepository

SUMMARY:
Prospective, observational registry for subjects with SLE under the care of a rheumatology provider. Longitudinal data are collected from both subjects and their treating rheumatology provider during routine clinical encounters using a structured and standardized data collection method.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of Systemic lupus erythematosus (SLE) subjects to evaluate long-term real-world safety and effectiveness of standard of care treatments for SLE. Data collected through the registry may be used to address a range of research questions and use cases, including but not limited to: characterizing the natural history of the disease, evaluating the effectiveness and safety of commercially available medications for the treatment of SLE, providing information to support ongoing risk-benefit evaluation by drug manufacturers and regulators, and research related to drug utilization, disease burden, and unmet needs. Further, data collected will inform clinical decision making by patients and treating providers. This will be enabled through the standardized data collection including validated patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization data.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this registry, an individual must meet all the following criteria:

1. Has been diagnosed with SLE by a rheumatologist or a qualified rheumatology practitioner.
2. Is at least 18 years of age or older and has attained the legal age for consent to procedures involved in the research, under the applicable law of the jurisdiction in which the research is being conducted at the time of enrollment.
3. Willing and able to provide informed consent.
4. Willing and able to provide Personally Identifiable Information (full legal name, sex at birth, date of birth, and home address zip/postal code at a minimum) if required based on registry location and applicable laws and regulations.
5. In addition, subjects must meet at least one of the following criteria:

   * New diagnosis of SLE (=<12 months) from registry enrollment, OR
   * Initiation of a biologic or immunosuppressant for the treatment of SLE at registry enrollment, OR
   * Lupus Nephritis (LN; class III-V) diagnosed within 2 years of registry enrollment

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in the registry:

1. Is participating in a double-blind clinical trial for a SLE drug
2. Subjects participating in any non-blinded trial for any indication, with the exception of non-blinded CAR-T or other cell/gene therapies for the treatment of SLE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled in the registry should be at least 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
SLE epidemiology and presentation, | Every 6 months for 10 years
  The major clinical outcome include an assessment of the epidemiology of Systemic Lupus Erythematosus; to better understand the presentation and natural history.
SLE management, and outcomes | Every 6 months for 10 years
  The major clinical outcome include an assessment of the epidemiology of Systemic Lupus Erythematosus; to better understand the management and outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, Waltham, Massachusetts, United States